CLINICAL TRIAL: NCT05707507
Title: Implementation of an Outpatient Parenteral Antimicrobial Therapy Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. Adrian Camacho-Ortiz, Head of Infectious Diseases Department, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IF22-00011
Record Dates: First submitted 2023-01-16; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Outpatient
Keywords: OPAT; Outpatient; Mexico

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient antimicrobial therapy (Active Comparator): Included patients will receive outpatient antimicrobial therapy according to their infectious disease.
  Interventions: Other: Place of treatment
- Inpatient antimicrobial therapy (Other): Included patients will receive intrahospital antimicrobial therapy according to their infectious disease.
  Interventions: Other: Place of treatment

INTERVENTIONS:
Other: Place of treatment — Patients with an infectious diseases have to be treated with a specify antimicrobial therapy. The differences between the arms is about the possibility to continue with the treatment in or out of the hospital.

SUMMARY:
To determine cost changes with an Outpatient Parenteral Antimicrobial Therapy Program (OPAT) treatment compared to standard therapy while maintaining safety and efficacy.

DETAILED DESCRIPTION:
Patients will be evaluated during the period January 2023 to January 2024. Patients over 18 years admitted to the University Hospital Dr. José Eleuterio González with microbiological diagnosis of an infection that needs an intravenous antimicrobial treatment for more than three days, without other criteria to remain hospitalized.

Informed consent will be provided to the patient, which is a requirement to enter the study, on it we will explain in detail the processes and follow-ups that you will have during participation in the study, as well as the confidentiality of personal data and results.

After signing informed consent, patients will be randomized 1:1 to enter the OPAT group or the inpatient antimicrobial therapy group.

Subjects will be stratified according to the diagnosed infection and will be followed within the protocol up to 30 after the end of the antimicrobial treatment established by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Infectious disease confirmed
* Need to be treated for 3 or more days
* Suitable catheter/venous access

Exclusion Criteria:

* Patients who have to be hospitalized for other cause
* Age < 18 years
* Pregnancy
* Not appropriate catheter/venous access
* Patients who changed of hospital
* Patients who got any other medical insurance
* Patients absent for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Cost changes with an Outpatient Parenteral Antimicrobial Therapy Program (OPAT) treatment compared to standard intrahospital therapy. | 1 year
  Total OPAT costs will be estimated from actual costs and readmissions costs after adverse events that would not have occurred if patients had been treated as inpatients.
  Actual costs will be obtained from the annual financial records of the service during the study period. These will include staff salaries, medications, equipment, and other costs.
  To estimate the costs of conventional care that would have been incurred if patients were treated as inpatients, it will be assumed that intrahospital stay would be equal to the OPAT care with the same diagnosis.

SECONDARY OUTCOMES:
Saved bed days | 1 year
  The bed days saved will be determined by calculating the number of days between the start and end of care at OPAT.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario José E. Gonzalez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Psaltikidis EM, Silva END, Moretti ML, Trabasso P, Stucchi RSB, Aoki FH, Cardoso LGO, Hofling CC, Bachur LF, Ponchet DDF, Colombrini MRC, Tozzi CS, Ramos RF, Costa SMQ, Resende MR. Cost-utility analysis of outpatient parenteral antimicrobial therapy (OPAT) in the Brazilian national health system. Expert Rev Pharmacoecon Outcomes Res. 2019 Jun;19(3):341-352. doi: 10.1080/14737167.2019.1541404. Epub 2018 Nov 5. PMID 30362845
- [Result] Seaton RA, Barr DA. Outpatient parenteral antibiotic therapy: principles and practice. Eur J Intern Med. 2013 Oct;24(7):617-23. doi: 10.1016/j.ejim.2013.03.014. Epub 2013 Apr 18. PMID 23602223
- [Result] Bernard L, El-Hajj, Pron B, Lotthe A, Gleizes V, Signoret F, Denormandie P, Gaillard JL, Perronne C. Outpatient parenteral antimicrobial therapy (OPAT) for the treatment of osteomyelitis: evaluation of efficacy, tolerance and cost. J Clin Pharm Ther. 2001 Dec;26(6):445-51. doi: 10.1046/j.1365-2710.2001.00380.x. PMID 11722682
- [Result] Amodeo MR, Clulow T, Lainchbury J, Murdoch DR, Gallagher K, Dyer A, Metcalf SL, Pithie AD, Chambers ST. Outpatient intravenous treatment for infective endocarditis: safety, effectiveness and one-year outcomes. J Infect. 2009 Dec;59(6):387-93. doi: 10.1016/j.jinf.2009.09.009. Epub 2009 Sep 17. PMID 19766136
- [Result] Durojaiye OC, Bell H, Andrews D, Ntziora F, Cartwright K. Clinical efficacy, cost analysis and patient acceptability of outpatient parenteral antibiotic therapy (OPAT): a decade of Sheffield (UK) OPAT service. Int J Antimicrob Agents. 2018 Jan;51(1):26-32. doi: 10.1016/j.ijantimicag.2017.03.016. Epub 2017 Jun 30. PMID 28673610